CLINICAL TRIAL: NCT00188097
Title: Diagnosis of Variceal Bleeding and Its Control in Cirrhosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PHRC 03-04
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2006-01-19 (Estimated); Status verified 2005-08

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

INTERVENTIONS:
Behavioral: Diagnosis of variceal bleeding and dits control in cirrhosis

SUMMARY:
The aim of the study was to determine the independent predictors of variceal bleeding and control of bleeding in cirrhosis as no scientific assessment have been perfomed until now

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients admitted for an acute complication of cirrhosis
* admission ≤ 6 hours of inclusion

Exclusion Criteria:

* Child-Pugh score > 13
* Digestive hemorrhage
* Non cirrhotic portal hypertension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 1999-11; Study Completion 2002-06

PRIMARY OUTCOMES:
variceal bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cales, PHD, Principal Investigator — UH Angers